CLINICAL TRIAL: NCT03985306
Title: Treatment of Diabetic Foot Ulcers With Inforatio Technique to Promote Wound Healing: a Feasibility Trial
Brief Title: Treatment of Diabetic Foot Ulcers With Inforatio Technique to Promote Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-122-2018
Record Dates: First submitted 2019-03-25; First posted 2019-06-13 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Wound Heal; Ulcer Foot; Ulcer Healing
Keywords: Diabetic foot ulcer; Wound treatment; Inforatio technique; Diabetes; Foot ulcer; Outpatient clinic; Feasibility trial; Punch biopsy; Foot ulcer treatment
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The trial is a single-center single-group feasibility trial in outpatient clinical settings.
  The trial will be reported with reference to the extended CONSORT guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility trial group (Experimental): Every trial patient will receive the intervention (the inforatio technique) that is intended for the definitive randomized clinical trial.
  Interventions: Procedure: Inforatio technique

INTERVENTIONS:
Procedure: Inforatio technique — We define the inforatio technique as punch biopsies taken in the periphery of the wound bed. The punch biopsies will have a diameter of two mms. The depth of the biopsies is primarily based on clinical assessment on distance to bone by assessment with a sterile wound probe and with attention to location and anatomy. The maximum depth will be 3.5 millimeters. The biopsies will be taken from one to two mms from the wound edges and with a distance of five mms between the biopsies.
  Inforatio technique is applied after standard care and wound assessment.

SUMMARY:
This trial will examine the feasibility of conducting a definitive randomized clinical trial that tests whether inforatio technique will reduce time to healing of diabetic foot ulcers. Inforatio technique is a procedure where small punch biopsies are taken from the wound bed near the edge of the wound. With this technique, the investigators wish to initiate an acute inflammatory response that increases the generation of granulation tissue with subsequent healing by scar formation. Thus, the investigators hypothesize that inforatio technique will promote healing of diabetic foot ulcers.

Based on clinical experience, the investigators have previously detected a reduction in time to healing as an unexpected effect when multiple punch biopsies are taken from the wound bed of diabetic foot ulcers. To the knowledge of the investigators, methods similar to the inforatio technique has not previously been studied.

DETAILED DESCRIPTION:
BACKGROUND

The prevalence of diabetic foot ulcers is expected to increase considerably due to a continuously increasing prevalence of diabetes. The healing process of diabetic foot ulcers is complicated by a complex pathophysiology of the distal lower extremities and a constant exposure to bacteria and pressure. Improving healing of diabetic foot ulcers will have several benefits including higher quality of life, reduced morbidity, reduced mortality and lower socioeconomic costs. Nonetheless, there are few randomized controlled clinical trials on surgical and non-surgical treatment chronic foot ulcers and many studies on the topic have a low level of evidence.

TRIAL AIMS

The investigators aim to assess the feasibility of conducting a definitive randomized controlled trial by exploring recruitment, patient acceptability, protocol adherence and adverse effects.

The success criteria of the trial is as follows:

* Weekly recruitment rates at two patients or more.
* Time from first outpatient visit to recruitment at 21 days or less.
* Retention rate at 90-day follow-up at 50% or more
* No appearance of unacceptable adverse effects In addition, the trial aims to assess logistic concerns regarding the trial and to improve the method of inforatio application.

Based on findings from the feasibility trial, the investigators may amend the design of the definitive trial.

RECRUITMENT

Patients are eligibility-screened and identified by the primary investigator and wound care staff when patients visit wound outpatient clinics at the recruiting facilities.

INCLUSION AND FOLLOW-UP

Eligible patients are included if they give their oral and written consent to participate. The baseline trial visit take place on the day that patients give their consent to participate.

The trial comprises a 90-day clinical follow-up. Follow-up visits will be at 10, 21, 42 and 90 days after baseline (give or take 3 days). Wounds are assessed at each trial visit. The inforatio technique is applied at baseline and again at the 21-follow-up day if the wound still has a diameter larger than four mms. Participants unable to attend at the precise dates for midtrial follow-up will be eligible for follow-up three days before or after the intended date. The participants who cannot attend during this window will skip the follow-up day in concern. If the participants miss the second intervention at the 21-day follow-up, they are excluded. For the 90-day follow-up, participants are recalled two times by the primary investigator within two weeks before being excluded.

Participants exit from the trial if following occurs during follow-up:

* they undergo surgeries described in the exclusion criteria
* they get acute signs of infection, gangrene or osteomyelitis in their foot in concern
* their tendons, joints or bone become exposed in the wound bed
* they develop an acute phase of charcot arthropathy in their foot in concern
* they get admitted for reasons related to their foot ulcer
* they die or emigrate

The trial is stopped if the intervention shows an unintended effect or potential harm.

TRIAL STANDARD TREATMENT

The participants receive a trial standard treatment at every trial visit. The treatment is conducted by the primary investigator in cooperation with wound care nurses and podiatrists. The standard treatment is defined based on Danish National guidelines, local guidelines of the recruiting facilities and guidelines of the National Institute for Health and Care Excellence.

The treatment is based on a flowchart that individualizes treatment based on clinical wound characteristics.

INFORATIO TECHNIQUE

The technique is described in the Arms and Interventions section.

TRIAL MEASURES

Wound assessment: Wounds are assessed at every trial visit. To monitor the ulcer area during follow-up, the investigators will analyze digital photos of the ulcer by using Image J which is a wound planimetry software. The depth of the ulcers are measured with sterile wound probes and reported by intervals of 5 millimeters. Undermining will be assessed with the same method as for depth and in intervals of 5 millimeters.

Microbial samples: At both stages of inforatio application, three punch biopsies are sent for cultivation to analyze bacterial species, bacterial load and resistance patterns of the bacteria.

Patient and staff interviews: described in the Outcome Measures section

STATISTICAL ANALYSIS

With descriptive statistics participants' demographics, the quantitative success criteria, the quantitative outcome measures and time to healing will be reported. Clinical healing is defined by intact epithelia.

The investigators will use statistical software SPSS version 21.0 (IBM Corp., Armonk, New York).

SAMPLE SIZE CONSIDERATION

Because effectiveness is not evaluated, a formal power calculation is not considered necessary for the objectives of a feasibility trial.

To minimize the number of patients that are exposed to a new intervention meanwhile keeping a level of precision for the variance estimate, the rule of thumb by Julious et al will be used for determination of the trial sample size. Thus, 12 participants will be included in the trial. Julious et al argues that a sample size of 12 per group gives a sufficient precision of the mean and variance estimates. Other studies report rules of thumbs with larger sample size to gain sufficient power for a pilot or feasibility trial.

ETHICAL CONSIDERATIONS AND RISK ASSESSMENT OF SIDE EFFECTS

The procedure of the intervention is small with an expectedly small risk of harm outcomes. The punch biopsies from the inforatio technique is relatively shallow therefore it is not expected that it will penetrate important anatomical structures or expose bone.

The primary investigator's clinical assessment, patient preference and patient tolerance is taken into consideration before inforatio technique is applied. Minimal discomfort is expected for the participants when they receive the inforatio technique treatment. Previous applications by the investigators showed that patients reported no or little pain during application.

The inforatio technique treatment has previously shown potential to improve healing thus participants may gain an improvement in healing of their foot ulcers.

If this trial shows that a definitive randomised clinical trial will be feasible, the investigators will examine the effect of inforatio technique through a larger randomised clinical trial. If the inforatio technique shows significant positive effect on time to healing it would become of great importance for future diabetic foot ulcer patients. The inforatio technique would become an addition to available therapeutic options. The technique is simple and only requires a punch biopsy tool. Nurses and general practitioners can be potential applicants that apply the treatment at clinics close to patient habitats making visits for wound treatment more convenient for the patients. If there is a significant positive effect on healing, it is expected that it will result in reduction of hospital admissions and less surgical interventions including amputations.

This project may contribute to more focus on treatment of patients with diabetic foot ulcers - a field of research that still needs studies to enable evidence-based treatment.

Inspectors from The National Committee of Health Research Ethics will have the authorization to quality control the trial.

COMPETING INTERESTS

The trial investigators declare that they have no competing interests.

ELIGIBILITY:
INCLUSION CRITERIA:

We include diabetic patients with foot ulcers that are more than six weeks old and which are located distal to the malleoli.

The diameters of the ulcers must be at least four mms. One wound from each foot of a patient can be included. If a patient's foot have more than one ulcer that meets the abovementioned criteria, the biggest wound is included. If there is no difference in size, the wound that has the most recent onset is included. If two wounds are close to each other and separated by less than 5 mm intact skin, we will consider it as one wound.

Wound onset estimates will be patient-reported.

EXCLUSION CRITERIA:

We exclude following patients:

* Patients with dementia and other patients who are not able to give their informed consent.
* Patients with gangrene, necrosis deeper than 1mm, osteomyelitis and clinical signs of infection in their foot. Infection is identified by clinical assessment based on the classical signs comprising oedema, pain, warmth, redness and purulent exudates and is assessed by an experienced orthopedic surgeon.
* Patients with ulcers that have positive probe-to-bone test and visible joint and tendons
* Patients with systolic toe pressure of < 20 mmHg
* Patients that, since the onset of their present foot ulcer, underwent vascular surgery in the lower extremity with the same laterality as the foot ulcer.
* Patients that, since the onset of their present foot ulcer, underwent surgical off-loading and amputations
* Patients that, since the onset of their present foot ulcer, underwent surgical wound revisions in an operating room.
* Patients that have an acute phase of Charcot arthropathy in the foot that presents with a foot ulcer.
* Patients that take systemic immunosuppressive drugs.
* Patients with cancer
* Patients with scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Eligibility rates | The first 2 months of the trial (untill the last patient has been recruited)
  Descriptive statistics of number and rate of eligible patients during the period of recruitment
Refusal rates | The first 2 months of the trial (untill the last patient has been recruited)
  Descriptive statistics of number and rate of eligible patients that refuse trial participation.
Time from identification to inclusion | The first 2 months of the trial (untill the last patient has been recruited)
  Descriptive statistics of average time from eligible patients are identified to they are included in the trial (baseline trial visit)
Qualitative assessment of unexpected factors that must cause exclusion | 10 months
  Qualitatively assessed by the primary investigator
Rate of unexpected exclusion | 10 months
  Descriptive statistics of number and rate of patients that are excluded due to reasons not already covered by the trial definition of exclusion criteria.
Retention rates | 10 months
  To investigate protocol adherence, the number and rate of participants that adhere to follow-up will be reported.
Number of missed trial follow-up visits | 10 months
  To investigate protocol adherence, the number of missed trial visits will be reported for each participant.
Drop-out rates | 10 months
  To investigate protocol adherence, the number and rate of participants that choose to drop out during follow-up will be reported.
Rate of eligible patients that accept participation | At baseline, each follow-up visit and when patients drop out.
  A quantitative investigation of patient acceptability.
Qualitative assessment of patient acceptability | 10 months
  Assessed by interviews with participants.
Observed harms and unexpected effects | 10 months
  Observed harms and unexpected effects observed by the investigators and staff will be reported.
Patient-reported potential side effects | 10 months
  A qualitatively assessment of harms and unexpected effects by interviewing participants about potential side effects that they experience.
Qualitative assessment of logistics issues regarding outpatient clinic visits | 10 months
  The investigators qualitatively assesses logistic circumstances that may be optimized.The assessment includes whether dates of follow-up visits fit the routines at the outpatient clinics.
Time to healing of punch biopsy scars | 10 months
  The time to healing will be reported to estimate if and when observer blinding may be possible.
Qualitative assessment of the method of wound assessment. | 10 months
  The investigators assess complications related to the method wound bed area and the depth. The aim is to optimize wound assessment for the future definitive trial.
Qualitative assessment of the extent of qualitative patient measures | 10 months
  The investigators assess whether the qualitative patient measures are either too extensive or insufficient. Thus, estimating necessary changes to make the qualitative measurements feasible to include in the future definitive trial.
Qualitative assessment of the feasibility of culturing 3 biopsies from each round of inforatio technique applications for a future definitive trial. | 10 months
  The investigators assess whether the included centers have the capacity to culture three biopsies two times from each patient.
Rates of wound treatments at trial visits that deviate from the trial standard treatment definition | 10 months
  Standard treatments received by each patient at the follow-up visits are recorded and it is assessed whether the standard care received corresponds to the definition of the trial standard treatment.
Qualitative assessment of wound care treatments received between trial visits and the deviations from the trial definition of standard treatment. | 10 months
  The investigators assess the heterogeneity of treatment during follow-up by recording the number of hospital visits between the trial follow-up visits and the treatments and assessments received at these hospital visits.
Time to healing of the foot ulcers | 10 months
  The investigators will report mean and variance of time to healing
Patient-reported experience of trial participation and the inforatio technique | 10 months
  The investigators will interview the patient about their experience of trial participation and of the inforatio technique.
Staff acceptability | 10 months
  Assessed qualitatively by interviews with the staff at the outpatient clinics (wound care nurses and podiatrists)
Qualitative assessment of the inforatio technique | 5 months. At baseline application and at the 21-day applications.
  The method of inforatio technique application will be qualitatively assessed by the applicant. The applicant will report any issues or complications regarding the inforatio technique definition.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Moeini, MD, Principal Investigator — Zealand University Hospital Koege, Denmark; Hans Gottlieb, Chief consultant, MD PhD, Study Chair — Herlev University Hospital, Denmark; Tue S Jørgensen, MD PhD, Study Chair — Hvidovre University Hospital, Denmark; Malene RB Larsen, MD, Study Chair — Zealand University Hospital Koege, Denmark; Stig Brorson, Professor, MD PhD DMsc, Principal Investigator — Zealand University Hospital Koege, Denmark
Locations (2):
- Denmark (2):
  - Herlev University Hospital, Department of Orthopaedic Surgery, Herlev
  - Zealand University Hospital, Department of Orthopaedic Surgery, Køge

REFERENCES:
- [Background] Andrews KL, Houdek MT, Kiemele LJ. Wound management of chronic diabetic foot ulcers: from the basics to regenerative medicine. Prosthet Orthot Int. 2015 Feb;39(1):29-39. doi: 10.1177/0309364614534296. PMID 25614499
- [Background] Karri VV, Kuppusamy G, Talluri SV, Yamjala K, Mannemala SS, Malayandi R. Current and emerging therapies in the management of diabetic foot ulcers. Curr Med Res Opin. 2016;32(3):519-42. doi: 10.1185/03007995.2015.1128888. Epub 2016 Jan 12. PMID 26643047
- [Background] Zimny S, Pfohl M. Healing times and prediction of wound healing in neuropathic diabetic foot ulcers: a prospective study. Exp Clin Endocrinol Diabetes. 2005 Feb;113(2):90-3. doi: 10.1055/s-2004-830537. PMID 15772900
- [Background] Greer N, Foman N, Dorrian J, Fitzgerald P, MacDonald R, Rutks I, Wilt T. Advanced Wound Care Therapies for Non-Healing Diabetic, Venous, and Arterial Ulcers: A Systematic Review [Internet]. Washington (DC): Department of Veterans Affairs (US); 2012 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK132238/ PMID 23586115
- [Background] Game FL, Apelqvist J, Attinger C, Hartemann A, Hinchliffe RJ, Londahl M, Price PE, Jeffcoate WJ; International Working Group on the Diabetic Foot. Effectiveness of interventions to enhance healing of chronic ulcers of the foot in diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:154-68. doi: 10.1002/dmrr.2707. PMID 26344936
- [Background] Braun LR, Fisk WA, Lev-Tov H, Kirsner RS, Isseroff RR. Diabetic foot ulcer: an evidence-based treatment update. Am J Clin Dermatol. 2014 Jul;15(3):267-81. doi: 10.1007/s40257-014-0081-9. PMID 24902659
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Braun L, Kim PJ, Margolis D, Peters EJ, Lavery LA; Wound Healing Society. What's new in the literature: an update of new research since the original WHS diabetic foot ulcer guidelines in 2006. Wound Repair Regen. 2014 Sep-Oct;22(5):594-604. doi: 10.1111/wrr.12220. PMID 25139424
- [Background] SIGN. 116 Management of diabetes. A national clinical guideline. 2017; Available from: https://www.sign.ac.uk/assets/sign116.pdf
- [Background] NICE Guideline. Diabetic foot problems: prevention and management [Internet]. [cited 2019 Jan 3]. Available from: https://www.nice.org.uk/guidance/ng19
- [Background] Rogers LC, Bevilacqua NJ, Armstrong DG, Andros G. Digital planimetry results in more accurate wound measurements: a comparison to standard ruler measurements. J Diabetes Sci Technol. 2010 Jul 1;4(4):799-802. doi: 10.1177/193229681000400405. PMID 20663440
- [Background] Schweitzer ME, Daffner RH, Weissman BN, Bennett DL, Blebea JS, Jacobson JA, Morrison WB, Resnik CS, Roberts CC, Rubin DA, Seeger LL, Taljanovic M, Wise JN, Payne WK. ACR Appropriateness Criteria on suspected osteomyelitis in patients with diabetes mellitus. J Am Coll Radiol. 2008 Aug;5(8):881-6. doi: 10.1016/j.jacr.2008.05.002. PMID 18657783
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharm Stat [Internet]. 2005;4(4):287-91. Available from: https://onlinelibrary.wiley.com/doi/abs/10.1002/pst.185
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] O'Meara SM, Cullum NA, Majid M, Sheldon TA. Systematic review of antimicrobial agents used for chronic wounds. Br J Surg. 2001 Jan;88(1):4-21. doi: 10.1046/j.1365-2168.2001.01631.x. PMID 11136304
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581